CLINICAL TRIAL: NCT06137092
Title: A Randomized, Two-armed, Double-blind, Single-dose, Crossover, Two-sequence, Bioequivalence Clinical Trial to Compare PK Parameters and Safety of rFVIII-Fc (AryoGen Pharmed Co.) Versus Elocta® in PTPs With Severe Hemophilia A
Brief Title: rFVIII-Fc (Produced by AryoGen Pharmed Co.) Pharmacokinetic Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AryoGen Pharmed Co. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FVIII.ARY.AE.00.PK
Record Dates: First submitted 2023-10-30; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-10

CONDITIONS: Severe Hemophilia A
MeSH Terms: conditions — Hemophilia A | interventions — Factor VIII

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AryoGen Pharmed Co. rFVIII-Fc/Elocta® (Sobi Co. rFVIII-Fc) (Experimental): AryoGen Pharmed Co. rFVIII-Fc, IV, 50 units/kg, single dose, then Elocta® (Sobi Co. rFVIII-Fc), IV, 50 units/kg, single dose (cross-over)
  Interventions: Drug: Factor VIII, recombinant human with Fc fusion (rFVIII-Fc)
- Elocta® (Sobi Co. rFVIII-Fc)/AryoGen Pharmed Co. rFVIII-Fc (Experimental): Elocta® (Sobi Co. rFVIII-Fc), IV, 50 units/kg, single dose, then AryoGen Pharmed Co. rFVIII-Fc, IV, 50 units/kg, single dose (cross-over)
  Interventions: Drug: Factor VIII, recombinant human with Fc fusion (rFVIII-Fc)

INTERVENTIONS:
Drug: Factor VIII, recombinant human with Fc fusion (rFVIII-Fc) — rFVIII-Fc, IV, 50 units/kg/ single dose, cross-over

SUMMARY:
The study is designed as a randomized, two-armed, double-blind, single-dose, crossover, two-sequence, active-controlled, multi-center, bioequivalence clinical trial with a primary endpoint of dose-normalized area under the curve (dnAUC last)

ELIGIBILITY:
Inclusion Criteria:

* Male patients ≥ 12 years, with signed informed consent by the patient, or the patient's legally authorized representative for patients under the legal age
* Diagnosed with severe hemophilia A (endogenous FVIII <1% [1 IU/dL])
* History of at least 150 documented prior exposure days to any FVIII product
* Having adequate bone marrow and organ function:

  * Plt ≥ 80,000 cells/µL
  * Hb ≥ 8 mg/dL
  * eGFR ≥ 30 mL/min
  * ALT or AST ≤ 5×ULN
  * Serum bilirubin ≤ 1.5×ULN

Exclusion Criteria:

* Measurable anti-drug antibody activity against FVIII (≥ 0.6 BU/mL) at screening or a history of developing anti FVIII antibody
* History of other coagulation disorders except for hemophilia A
* Acute hemorrhagic state
* Infection with HCV or HBV
* HIV-positive patients
* Infusion of any products containing FVIII within 7 days prior to first administration
* Previous treatment with commercially available extended half-life FVIII products
* Receiving drugs which increase bleeding tendency (e.g: Anti-coagulants, antiplatelets, omega 3, Vit E, etc.) within 2 weeks of screening. NSAIDs are permitted.
* Current systemic treatment with immunosuppressive drugs
* Hypersensitivity or anaphylaxis associated with any FVIII concentrate or intravenous immunoglobulin (IVIG)
* Planned elective surgery
* Current enrolment or willing to enroll in any other experimental study during the time of current trial
* Subjects assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol (e.g.: physical, psychological and mental problems)

Min Age: 12 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Only male patients are eligible for the study.
Enrollment: 50 (Actual)
Dates: Start 2023-07-22 (Actual); Primary Completion 2023-09-27 (Actual); Study Completion 2023-09-27 (Actual)

PRIMARY OUTCOMES:
dose-normalized Area Under the Curve (dnAUC last) | pre-dose, 15 minutes, 30 minutes, 1 hour, 3 hours, 6 hours, 8 hours, 24 hours, 48 hours, 72 hours, 96 hours, 120 hours post-dose
  Area under the concentration-time curve measured from the time of administration to the last measurable time point

SECONDARY OUTCOMES:
Area Under the Curve to Infinity (AUC inf) | pre-dose, 15 minutes, 30 minutes, 1 hour, 3 hours, 6 hours, 8 hours, 24 hours, 48 hours, 72 hours, 96 hours, 120 hours post-dose
  Area under the concentration-time curve measured from the time of administration to the infinity.
Maximum Plasma Activity (Cmax) | pre-dose, 15 minutes, 30 minutes, 1 hour, 3 hours, 6 hours, 8 hours, 24 hours, 48 hours, 72 hours, 96 hours, 120 hours post-dose
  Maximum plasma activity during a dosing interval
Incremental Recovery (IR) | pre-dose, 15 minutes, 30 minutes, 1 hour
  The rise in FVIII activity in IU/dL per unit dose administered in IU/kg
Half-life (T ½) | pre-dose, 15 minutes, 30 minutes, 1 hour, 3 hours, 6 hours, 8 hours, 24 hours, 48 hours, 72 hours, 96 hours, 120 hours post-dose
  Time required for the activity of the drug to reach half of its original value
Volume of distribution (Vd) | pre-dose, 15 minutes, 30 minutes, 1 hour, 3 hours, 6 hours, 8 hours, 24 hours, 48 hours, 72 hours, 96 hours, 120 hours post-dose
  Volume of distribution estimated from the terminal phase
Clearance (Cl) | pre-dose, 15 minutes, 30 minutes, 1 hour, 3 hours, 6 hours, 8 hours, 24 hours, 48 hours, 72 hours, 96 hours, 120 hours post-dose
  Rate at which the body removes the drug, measured as the volume of the plasma cleared of drug per unit time per unit weight
Safety assessment by evaluation of adverse events (AEs) and abnormal laboratory results | Adverse events collection and documentation was done during the study (up to 28 days)
  Safety assessment, including the incidence of all reported AEs and abnormal laboratory results was done. All AEs were classified based on the Medical Dictionary for Regulatory Activities (MedDRA Desktop Browser 4.0 Beta) terms as System Organ Class (SOC) and Preferred Term (PT). All the reported events were graded according to the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0). Moreover, seriousness of AEs was assessed according to International Council for Harmonization (ICH-E2B) guidelines. The causality relation was assessed based on the World Health Organization (WHO) criteria.
Immunogenicity assessment | Immunogenicity sampling was done at screening visit and day 7, 12 and 28
  Immunogenicity of factor viii was evaluated at scheduled visits by blood sampling to determine the production of inhibitor against factor viii.

CONTACTS AND LOCATIONS:
Overall Officials: Aziz Eghbali, Assoc. Prof., Principal Investigator — Iran University of Medical Sciences
Locations (5):
- Iran (5):
  - Seyed-Al-Shohada Hospital, Isfahan
  - Sarvar Clinic, Mashhad
  - Dastqeib Hospital, Shiraz
  - Imam Khomeini, Tehran
  - Mofid Hospital, Tehran

REFERENCES:
- [Derived] Eghbali A, Eshghi P, Toogeh G, Alavi S, Badiei Z, Ghanavat M, Bordbar M, Bazrafshan A, Karimi K, Ahmadinejad M, Sabzvari A, Kafi H. A randomized, two-armed, double-blind, single-dose, cross-over, bioequivalence clinical trial to compare pharmacokinetic parameters and safety of recombinant human factor VIII with Fc fusion produced by AryoGen Pharmed Company versus Elocta(R) (reference product) in previously treated patients with severe haemophilia A. Ann Hematol. 2025 Feb;104(2):1195-1202. doi: 10.1007/s00277-025-06242-z. Epub 2025 Feb 12. PMID 39934428